CLINICAL TRIAL: NCT05805683
Title: Effect of Early Calcitonin Therapy on Incidence and Severity of Neuropathic Pain After Spinal Cord Injury
Brief Title: Calcitonin Therapy on Incidence and Severity of Neuropathic Pain After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, lecturer of anesthesiology, surgical intensive care and pain medicine Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 36264PR152/3/23
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-03

CONDITIONS: Calcitonin; Neuropathic Pain; Spinal Cord Injury
Keywords: Calcitonin; Neuropathic pain; Spinal cord injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries | interventions — Calcitonin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcitonin group (Experimental): patients in this group will receive 100 IU (1 ml) of calcitonin subcutaneously per day for 2 weeks starting within 48 hours after injury.
  Interventions: Drug: Calcitonin
- Placebo group (Placebo Comparator): patients in this group will receive 1 ml of saline placebo solution subcutaneously per day for 2 weeks starting within 48 hours after injury.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Calcitonin — patients in this group will receive 100 IU (1 ml) of calcitonin subcutaneously per day for 2 weeks starting within 48 hours after injury.
  Arms: Calcitonin group
Drug: Placebo — patients in this group will receive 1 ml of saline placebo solution subcutaneously per day for 2 weeks starting within 48 hours after injury.
  Arms: Placebo group

SUMMARY:
This prospective randomized double blinded study will be conducted to evaluate the effect of early pharmacologic intervention with calcitonin on the incidence or the severity of neuropathic pain after spinal cord injury

DETAILED DESCRIPTION:
Pain after spinal cord injury can be classified into five categories: musculoskeletal, visceral, at-level, above-level, and below-level neuropathic pain. Calcitonin has previously been shown to be effective in the management of acute pain following amputation, vertebral fractures and other neuropathic conditions. Also it was used in a previous study to prevent complex regional pain syndrome in severe hemiplegic patients after stroke

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years, with spinal cord injury at any level and any degree of completeness in the early stage of trauma.

Exclusion Criteria:

* Intake of anticonvulsants medications.
* Evidence of neuropathic pain.
* Evidence of previous allergic reaction to calcitonin.
* Patients with renal, hepatic and cardiac dysfunction or neurological disorders .
* brain damage or major trauma to extremities or abdomen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of neuropathic pain | 6 months after spinal cord injury
  Intensity of neuropathic pain will be evaluated by visual analogue scale (VAS) scores within the 1st 6 months after spinal cord injury
Incidence of chronic pain | 12 months after spinal cord injury
  Incidence of chronic pain at 12 months after spinal cord injury

SECONDARY OUTCOMES:
Incidence of neuropathic pain | 12 months after spinal cord injury
  Incidence of neuropathic pain at 1, 3, 6, 9 and 12 months after spinal cord injury
The incidence of adverse reactions | 2 weeks after spinal cord injury
  Nausea, vomiting, disturbance of serum Calcium, Magnesium and Phosphorus levels
The consumption of medications for neuropathic pain or musculoskeletal pain | 12 months after spinal cord injury
  Number of patients required medications for neuropathic pain or musculoskeletal pain
Intensity of neuropathic pain | 12 months after spinal cord injury
  Intensity of neuropathic pain will be evaluated by the visual analogue scale (VAS) score which ranges from 0 = no pain to 10= worst pain at 12 months after spinal cord injury
Intensity of nociceptive pain | 12 months after spinal cord injury
  Intensity of musculoskeletal pain will be evaluated by visual analogue scale (VAS) score which ranges from 0 = no pain to 10= worst pain at 1, 3, 6, 9 and 12 months after spinal cord injury

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available upon a reasonable request from the corresponding author after the end of study for 1 year
Access Criteria: The data will be available upon a reasonable request from the corresponding author